CLINICAL TRIAL: NCT06693479
Title: Could a Feedback Device Help Manage Work-related Shoulder Disorders? - Protocol of a Mixed Methods Pilot Study
Brief Title: Could a Feedback Device Help Manage Work-related Shoulder Disorders?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: The Arthritis Society, Canada (Other)
Responsible Party: Principal Investigator, Jean-Sébastien Roy, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MP-13-2023-2784
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Rotator Cuff-related Shoulder Pain; Shoulder Osteoarthritis; Rheumatoid Arthritis (RA)
Keywords: Technology; Shoulder pain; Feasibility; Workers; Feedback; Pilot; Randomized controlled trial; Focus group; Device; Mixed methods study
MeSH Terms: conditions — Arthritis, Rheumatoid; Shoulder Pain | interventions — Educational Status

STUDY DESIGN:
Masking Description: Due to the nature of the intervention, neither the treating physiotherapist nor the participants can be blinded. Blinding of the evaluator is irrelevant as outcome data will either be collected online with self-reported questionnaires or by the device measuring physical work demands. The investigator and statistician will remain unaware of group assignments throughout.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Device + Education (Experimental): Education session at week 2 and feedback from SWL during week 2 and week 3
  Interventions: Device: Shoulder watch load (SWL) feedback; Other: Education
- Education (Active Comparator): Education session at week 2.
  Interventions: Other: Education

INTERVENTIONS:
Device: Shoulder watch load (SWL) feedback — During week 2 and 3 after randomization, the experimental group will undergo the intervention using the SWL, designed to monitor workers' physical work demands. During this time, the SWL will provide real-time feedback based on parameters set via Ergowatchapp. A workplace visit by a physiotherapist will be conducted to establish and adjust the feedback thresholds in week 2, after the education intervention. If necessary, a second remote meeting will take place in week 3 to explain how participants can modify the thresholds themselves. The initial feedback thresholds will be set based on the physical work demands measured during week 1 and will be adjusted after one week of feedback use. These thresholds will be collaboratively determined by a physiotherapist and the workers. Only the experimental group will receive feedback from the SWL during the study period.
  Arms: Device + Education
Other: Education — Participants will receive an education intervention delivered by a physiotherapist. This intervention will take place preferentially at the participants' workplace at the end of the 2nd week post-randomization. The session will last 30 to 45 minutes, and involve personalized, patient-centered education on their condition. The physiotherapist will use open-ended questions to encourage participants to express their goals and address specific concerns related to their shoulder condition. Given the expected diversity in physical constraints (manual vs. non-manual workers) and individual challenges, the session will be tailored to each worker needs. At the end of the session, workers will receive a booklet summarizing key points, including: understanding shoulder anatomy, function and pain, managing shoulder pain, enhancing movement variability, adjusting work environment, and considering factors such as sleep, stress, coping mechanisms, and psychological factors on pain.

SUMMARY:
Work-related shoulder pain is a common problem with significant socio-economic repercussions. The impact of these disorders on workers is considerable, particularly in terms of pain, disability and reduced quality of life. Several occupational factors may explain the onset of these disorders, such as changes in the work environment, physical demands, psychosocial factors specific to the occupational context and the age of workers. The lack of quantitative measurement tools to assess the physical demands of work over an extended period of time is sorely felt. Recently, our team developed a wearable feedback device, similar to a watch worn on the arm, which measures shoulder movements and muscle activity, transforming this real-time data into clinical indicators. These indicators provide immediate feedback to workers, enabling them to better understand the physical demands of their tasks and adapt accordingly. If this device proves effective in reducing physical demands, it could become a valuable tool for guiding workplace assessments and interventions. However, this device has not yet been tested on workers with shoulder pain. For this reason, a two-part pilot study is needed to understand user needs, assess ease of use and the feasibility of implementing the device. The first component will consist of a pilot clinical trial involving 42 workers suffering from shoulder pain, divided into two groups: one group will use the feedback device for 2 weeks, while the other group will continue to work without intervention. The second phase will analyze the experience of participants who have used the device.

DETAILED DESCRIPTION:
The objectives of this pilot study are (a) to evaluate the feasibility of implementing the SWL in the workplace and conducting a large-scale randomized clinical trial (RCT) by assessing recruitment success, intervention adherence, acceptability of the technology, the research team's capacity to refine the SWL, and (b) to explore the SWL capacity to reduce disability, pain, work limitations, and physical work demands while increasing pain self-efficacy among workers with WRSDs.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≧ 18 years) employed full-time (minimum of 30 hours per week).
2. Experiencing work-related shoulder disorders (WRSDs), with minimal score of 14 points on the for the abbreviated version of the Disability of the Arm Shoulder and Hand questionnaire (QuickDASH), stemming from a diagnosis of rotator cuff-related shoulder pain (RCRSP), shoulder osteoarthritis (SOA) or rheumatoid arthritis (RA) involving the shoulder.
3. Symptoms persisting for more than 6 weeks.

Diagnosis-specific criteria:

1. RCRSP: diagnosis requires meeting three positive criteria, including the presence of a painful arc in abduction, a positive Neer sign, Hawkins-Kennedy test, or Jobe Test, pain with resisted humeral external rotation;
2. SOA: diagnosis based on clinical findings (e.g., activity-related pain, reduced range of motion particularly external rotation and function, worsening night/rest pain) and radiologic findings (e.g., osteophytes, joint space narrowing, subchondral sclerosis, cyst formations, and humeral head deformities);
3. RA involving the shoulder: confirmed diagnosis according to the American College of Rheumatology criteria.

Both SOA and RA diagnoses will be confirmed by a physician.

Exclusion Criteria:

1. clinical signs of a massive rotator cuff tear (e.g., pseudoparesis or pseudoparalysis, passive elevation intact but active limited to <90°, without neurologic deficit);
2. acute traumatic rotator cuff tears, fractures, adhesive capsulitis (characterized by night pain, pain with sudden or unexpected movements, global loss of active and passive range of motion), or shoulder instability (evidenced by a combination of orthopaedic tests such as apprehension and relocation tests, Jerk, Kim and posterior tests, along with and clinical signs like neuromuscular function impairment, history of instability, lesion mechanisms, worries that their shoulder could dislocate during activities);
3. distal neurovascular symptoms (e.g., thoracic outlet syndrome, venous thromboembolism);
4. previous shoulder surgery;
5. corticosteroid injection administered within the past 3 months;
6. symptomatic acromioclavicular joint pathology;
7. currently receiving conservative management for their shoulder pain (excluding medication for RA and OA),
8. absenteeism from work (unable to work at least 30 hours per week or on sick leave).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility : quantitative component procedure | Baseline
  Assessing trial recruitment success (Recruitment rate) : Track the rate of screened participants who consent to participate in the trial, using a screening and recruitment log.
Feasibility : quantitative component procedure | From enrollment to the end of recruitment
  Assessing trial recruitment success (Determining recruitment duration) : Evaluate the time required to recruit the target number of participants.
Feasibility : quantitative component procedure | From enrollment to the end the trial at 12 weeks
  Assessing trial recruitment success (Retention rate) : Monitor the number of participants who complete the trial, and document reasons for attrition.
Feasibility : quantitative component procedure | From enrollment to the end of the last completion questionnaire at 12 weeks
  Completion rate : Report the completion rate for each questionnaire at each time point.
Feasibility : quantitative component procedure | From 2 weeks to 4 weeks of the intervention period
  Evaluating adherence to the intervention : Self-reported SWL devise usage: Participants in the experimental group will complete a self-reported questionnaire at the end of each week during the 2-week intervention period to assess their adherence to using the SWL.
Feasibility : qualitative component procedure | From 4 weeks to 12 weeks
  Focus groups : All participants from the experimental group will be invited to participate to a focus group, to explore various aspects of feasibility such as the acceptability of the technology, the experience of wearing the SWL and receiving the feedback, and suggestion for potential improvement of the SWL.

SECONDARY OUTCOMES:
Abbreviated version of the Disability of the Arm Shoulder and Hand questionnaire-Work Module (QuickDASH-Work Module) | Baseline, 3 weeks, 6 weeks, 12 weeks
  QuickDASH-Work Module includes 4 items, each scored from 1 to 5. This scale range from 0 to 100, with 0 indicating the best function and 100 indicating the worst possible function
Abbreviated version of the Disability of the Arm Shoulder and Hand questionnaire (QuickDASH) | Baseline, 3 weeks, 6 weeks, 12 weeks
  The QuickDASH consists of 11 items, , each scored from 1 to 5. This scale range from 0 to 100, with 0 indicating the best function and 100 indicating the worst possible function.
Work Limitations Questionnaire (WLQ-25). | Baseline, 3 weeks, 6 weeks, 12 weeks
  This 25-item questionnaire includes four subscales addressing four dimensions of job demands. The total score ranges from 0 to 100, with 0 indicating no limitation and 100 indicating complete limitation
Pain severity subscale of the Brief Pain Inventory Short Form (BPI-SF) | Baseline, 3 weeks, 6 weeks, 12 weeks
  It includes 4 items measuring worst, least and average pain in the past 24 hours, as well as current pain, each scored on an 11-point numeric scale (0-10), where 0 indicates no pain and 10 represents the worst pain imaginable.
Pain Self-Efficacy Questionnaire (PSEQ). | Baseline, 3 weeks, 6 weeks, 12 weeks
  This questionnaire includes 10 items, each scored on a 7-point Likert scale (0 = not at all confident and 6 = completely confident).
Western Ontario Rotator Cuff Index (WORC) | Baseline, 3 weeks, 6 weeks, 12 weeks
  The WORC contains 21 items in total, each scored from 0 to 100, with 0 indicates best function and 100 indicating the worst possible function.
Physical work demands | At 1 week and 4 weeks
  To evaluate physical work demands, workers in both groups will wear the SWL for three consecutive full working days during the 1st week (before the intervention for the experimental group). Participants will log their physical work demands daily using the Ergowatchapp via a Mycap entry. The following outcomes will be averaged for data analysis: 1) number of arm elevations (>60°) per day, 2) time spent with the arm elevated (>60°) per day.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Meidinger, PT, PhD student, PT, PhD student, Principal Investigator — Centre interdisciplinaire de recherche en réadaptation et intégration sociale (Cirris); Jean-Sébastien Roy PT, PhD, Study Director — Centre interdisciplinaire de recherche en réadaptation et intégration sociale (Cirris)
Locations (1):
- Centre interdisciplinaire de recherche en réadaptation et intégration sociale (Cirris), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication (with anonymized data).
Time Frame: All data will be available starting after 6 months after publication (with anonymized data).
Access Criteria: For further information, please contact the authors

REFERENCES:
- [Derived] Meidinger P, Hong QN, Tittley J, Campeau-Lecours A, Roy JS. Could a feedback device help manage work-related shoulder disorders?: protocol of a mixed methods pilot study. Pilot Feasibility Stud. 2025 Jun 20;11(1):84. doi: 10.1186/s40814-025-01646-0. PMID 40542393
- See also: Could a feedback device help manage work-related shoulder disorders? - Protocol of a mixed methods pilot study — https://www.researchsquare.com/article/rs-5183538/v1